CLINICAL TRIAL: NCT04242420
Title: Impact of Connexin 37, Connexin 43 on Clinical Disease Phenotype in Delta F508 Homozygous Patients With Cystic Fibrosis (CF) (CF-Modifier)
Brief Title: Connexin Genotypes in Cystic Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Childrens' Hospital (Zentrum für Kinderheilkunde des Universitätsklinikum Bonn) (Other)
Collaborators: Goethe University (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Sabina Schmitt-Grohe, Principal investigator, University Childrens' Hospital (Zentrum für Kinderheilkunde des Universitätsklinikum Bonn)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BN 178/01
Record Dates: First submitted 2019-12-20; First posted 2020-01-27 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis; Inflammation
Keywords: connexin 37+43, MBL, TGF beta; Lung function; Interleukin 8
MeSH Terms: conditions — Cystic Fibrosis; Inflammation; Camurati-Engelmann Syndrome | interventions — Genotype; Respiration; Attachment Sites, Microbiological; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Evaluation of clinical parameters by genotype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connexin genotype (Other): Genotyping
  Interventions: Diagnostic Test: Genotyping; Diagnostic Test: Lung function; Diagnostic Test: Microbiology; Diagnostic Test: Blood sample; Diagnostic Test: Induced Sputum

INTERVENTIONS:
Diagnostic Test: Genotyping — Genotyping for single nucleotide polymorphisms for Connexin 37&43, Mannose binding lectin (MBL) and transforming growth factor beta (TGF beta) genotypes
Diagnostic Test: Lung function — Spirometry,
Diagnostic Test: Microbiology — Bacterial culture from Sputum or swab
Diagnostic Test: Blood sample — Interleukin-8 assay (via chemiluminescence) blood cell count
Diagnostic Test: Induced Sputum — Interleukin-8 assay (via chemiluminescence) blood cell count

SUMMARY:
Background: There is wide variety in lung disease phenotype for the delta F508 (homozygous) genotype. A leukocyte driven inflammation is most important for the pathogenesis of pulmonary disease in CF. Blood cytokines correlate negatively with pulmonary function in delta F508 homozygous patients. Gap junction proteins might be of importance for the influx of blood cells into the lung and may influence the course of pulmonary inflammation. A primary analysis (Horn et al. 2020) has shown that GJA4 variants (rs41266431) are linked to more severe disease in CF. This is very similar to variants of MBL.

Aims: To assess the relationship between gap junction proteins alpha 1 (GJA1/Connexin 43) and alpha 4 (GJA4/connexin 37) genotypes and clinical disease phenotype. Moreover are GJA4 variants in terms of clinical phenotype independent of MBL variants.

Methods:Patients homozygous for delta F508 get recruited from the CF centres of Bonn, Frankfurt and Amsterdam. Sequence analysis is performed for connexin 43 and 37 and MBL genotypes. Clinical disease is assessed longitudinally over 3 years by pulmonary function tests (FEV1 (forced expiratory volume in one second), FVC (=(forced vital capacity), FEF75 % (Forced expiratory flow at 75% of the pulmonary volume) pred), BMI (percentiles), P. aeruginosa colonization, diabetes mellitus and survival to end-stage CF lung disease (death or lung transplantation).

DETAILED DESCRIPTION:
Progressive pulmonary destruction is the major cause of morbidity and mortality in human subjects with cystic fibrosis. Many studies could not find an association between delta F 508 and severity of pulmonary disease . The most important factor in CF lung disease is an inflammation driven by leukocytes and cytokines. The investigators have provided evidence in former studies that cytokines (Interleukin-8 (IL-8), tumour necrosis factor (TNF) alpha, Lipopolysaccahride binding protein (LBP), transforming growth factor (TGF) ß)measured in blood correlate negatively with lung function in delta 508 homozygous patients.

The question arises, what other factors influence recruitment of proinflammatory leukocytes from blood capillaries into the lung .

Connexins are a family of transmembrane proteins, which oligomerize into hexameric structures to form a hemichannel (connexon) and ultimately pair with a partner hemichannel in an adjacent cell to form gap junction intercellular communication channels (GJIC) . There is evidence of expression of connexin 37 (=gap junction protein A4 (GJA4)) on macrophages in humans. Moreover there is evidence of expression of connexin 37 on vascular endothelia in humans . Connexin 37 is expressed on human neutrophils . Pulmonary disease in CF is dominated by a leukocyte driven inflammation. GAP junction proteins might be of importance for the influx of blood cells into the lung. In this regard, the hypothesis was that Cx37 or Cx43 genotypes have an impact on clinical disease phenotype in CF patients homozygous for delta F508. The first analysis (Horn et al 2020) has shown a clinical phenotype linked to the GJA4 genotype is very similar to MBL variants. In this regard the question arises whether there is a link between the MBL variant alleles and the GJA4 variants. Moreover some TGFbeta genotypes are linked to certain pulmonary phenotypes. So we are looking for interactions between Cx37 and TGFbeta genotypes and their impact on the clinical phenotype as well.

ELIGIBILITY:
Inclusion Criteria:

Homozygosity for delta F 508

Exclusion Criteria:

treatment with systemic steroids 14 days preceding this trial, participation in another study within the past 30 days, treatment with Orkambi or status after lung transplantation (for assessment of all parameters except survival).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2002-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival to end stage lung disease | through study completion, on average 27 years
  End stage lung disease: Death or lung transplantation
Lung function parameter: FEV1 | 3 years
  Best FEV1 value in % predicted of the year according to German registry according to Global lung initiative (GLI)
Lung function parameters: FVC | 3 years
  Best FVC value in % predicted of the year according to German registry according to Global lung initiative (GLI)
Lung function parameters: FEF75 | 3 years
  Best FEF75 value in % predicted of the year according to German registry according to Global lung initiative (GLI)

SECONDARY OUTCOMES:
Interleukin-8 in blood | through study completion, an average of 3 year
  single spot value (cross-sectional)
Interleukin-8 in sputum | through study completion, an average of 3 year
  single spot value (cross-sectional)
White blood cell count | through study completion, an average of 3 year
  Leukocytes (single spot value (cross-sectional))
Inflammatory markers in sputum | through study completion, an average of 3 year
  Leukocyte count in sputum (single spot value (cross-sectional))

OTHER OUTCOMES:
Colonisation with Pseudomonas aeruginosa | 3 years
  Never, Intermittent or chronic according to Leeds criteria
CF related diabetes mellitus | through study completion, an average of 3 year
  Assessment via patient charts/ registry

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Schmitt-Grohe, MD, Principal Investigator — University Hospital, Bonn
Locations (3):
- Germany (2):
  - University Hospital, Frankfurt, Hessia
  - University Hospital, Bonn, Nordrhine-Westphalia
- University Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drumm ML, Konstan MW, Schluchter MD, Handler A, Pace R, Zou F, Zariwala M, Fargo D, Xu A, Dunn JM, Darrah RJ, Dorfman R, Sandford AJ, Corey M, Zielenski J, Durie P, Goddard K, Yankaskas JR, Wright FA, Knowles MR; Gene Modifier Study Group. Genetic modifiers of lung disease in cystic fibrosis. N Engl J Med. 2005 Oct 6;353(14):1443-53. doi: 10.1056/NEJMoa051469. PMID 16207846
- [Result] Cystic Fibrosis Genotype-Phenotype Consortium. Correlation between genotype and phenotype in patients with cystic fibrosis. N Engl J Med. 1993 Oct 28;329(18):1308-13. doi: 10.1056/NEJM199310283291804. PMID 8166795
- [Result] McKone EF, Goss CH, Aitken ML. CFTR genotype as a predictor of prognosis in cystic fibrosis. Chest. 2006 Nov;130(5):1441-7. doi: 10.1378/chest.130.5.1441. PMID 17099022
- [Result] Schmitt-Grohe S, Naujoks C, Bargon J, Wagner TO, Schubert R, Hippe V, Zielen S. Interleukin-8 in whole blood and clinical status in cystic fibrosis. Cytokine. 2005 Jan 7;29(1):18-23. doi: 10.1016/j.cyto.2004.09.004. PMID 15579374
- [Result] Schmitt-Grohe S, Hippe V, Igel M, von Bergmann K, Posselt HG, Krahl A, Smaczny C, Wagner TO, Nikolazik W, Schubert R, Lentze MJ, Zielen S. Lipopolysaccharide binding protein, cytokine production in whole blood, and lipoproteins in cystic fibrosis. Pediatr Res. 2005 Nov;58(5):903-7. doi: 10.1203/01.PDR.0000182598.98167.24. Epub 2005 Sep 23. PMID 16183806
- [Result] Schmitt-Grohe S, Stuber F, Book M, Bargon J, Wagner TO, Naujoks C, Schubert R, Lentze MJ, Zielen S. TNF-alpha promoter polymorphism in relation to TNF-alpha production and clinical status in cystic fibrosis. Lung. 2006 Mar-Apr;184(2):99-104. doi: 10.1007/s00408-005-2568-x. PMID 16622779
- [Result] Eickmeier O, Boom Lv, Schreiner F, Lentze MJ, NGampolo D, Schubert R, Zielen S, Schmitt-Grohe S. Transforming growth factor beta1 genotypes in relation to TGFbeta1, interleukin-8, and tumor necrosis factor alpha in induced sputum and blood in cystic fibrosis. Mediators Inflamm. 2013;2013:913135. doi: 10.1155/2013/913135. Epub 2013 Aug 26. PMID 24062613
- [Result] Dempsie Y, Martin P, Upton PD. Connexin-mediated regulation of the pulmonary vasculature. Biochem Soc Trans. 2015 Jun;43(3):524-9. doi: 10.1042/BST20150030. PMID 26009202
- [Result] Chanson M, Derouette JP, Roth I, Foglia B, Scerri I, Dudez T, Kwak BR. Gap junctional communication in tissue inflammation and repair. Biochim Biophys Acta. 2005 Jun 10;1711(2):197-207. doi: 10.1016/j.bbamem.2004.10.005. Epub 2004 Oct 30. PMID 15955304
- [Result] Kwak BR, Mulhaupt F, Veillard N, Gros DB, Mach F. Altered pattern of vascular connexin expression in atherosclerotic plaques. Arterioscler Thromb Vasc Biol. 2002 Feb 1;22(2):225-30. doi: 10.1161/hq0102.104125. PMID 11834520
- [Result] Zahler S, Hoffmann A, Gloe T, Pohl U. Gap-junctional coupling between neutrophils and endothelial cells: a novel modulator of transendothelial migration. J Leukoc Biol. 2003 Jan;73(1):118-26. doi: 10.1189/jlb.0402184. PMID 12525569
- [Result] Saez PJ, Shoji KF, Aguirre A, Saez JC. Regulation of hemichannels and gap junction channels by cytokines in antigen-presenting cells. Mediators Inflamm. 2014;2014:742734. doi: 10.1155/2014/742734. Epub 2014 Sep 9. PMID 25301274
- [Result] Horn T, Ludwig M, Eickmeier O, Neerinex AH, Maitland-van der Zee AH, Smaczny C, Wagner TOF, Schubert R, Zielen S, Majoor C, Bos LD, Schmitt-Grohe S. Impact of a Gap Junction Protein Alpha 4 Variant on Clinical Disease Phenotype in F508del Homozygous Patients With Cystic Fibrosis. Front Genet. 2020 Oct 28;11:570403. doi: 10.3389/fgene.2020.570403. eCollection 2020. PMID 33193670
- [Derived] Laubach JP, Ludwig M, Horn T, Eickmeier O, Smaczny C, Schubert R, Zielen S, Majoor C, Aydin M, Schnell A, Schmitt-Grohe S. Transforming Growth Factor ss1 and Gap Junction Protein Alpha 4 Gene Heterogeneity in Relation to the Severity of Clinical Disease in Cystic Fibrosis. Front Biosci (Landmark Ed). 2023 Jul 19;28(7):138. doi: 10.31083/j.fbl2807138. PMID 37525914